CLINICAL TRIAL: NCT05312593
Title: Domiciliary Use of Hyaluronic Acid Gel Solutions vs Domiciliary Use of Chlorhexidine Mouthwash 0,20% for the Management of Peri-implant Mucositis Sites: a Randomized Clinical Trial
Brief Title: Domiciliary Use of Hyaluronic Acid Gel Solutions vs Domiciliary Use of Chlorhexidine Mouthwash 0,20% for the Management of Peri-implant Mucositis Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022-AFTORAL IMPL
Record Dates: First submitted 2022-03-26; First posted 2022-04-05 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Peri-implant Mucositis
Keywords: hyaluronic acid; chrlorhexidine; non-surgical periodontal therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial Group (Experimental): A group of 30 patients will be randomly assigned to Hyaluronic Acid domiciliary treatment, applied into Peri-implant mucositis sites.
  Interventions: Other: Aftoral Oral Gel
- Control Group (Active Comparator): A group of 30 patients will be randomly assigned to Chlorhexidine mouthwash domiciliary treatment, applied into Peri-implant mucositis sites.
  Interventions: Other: Unidea Chlorhexidine mouthwash

INTERVENTIONS:
Other: Aftoral Oral Gel — Patients will use Aftoral® Oral Gel solution for the domiciliary application once a day for 15 days after the visits (no rinsing and eating for 30 minutes after gel solution application).
  Arms: Trial Group
Other: Unidea Chlorhexidine mouthwash — Patients will use chlorhexidine mouthwash 0,20% for the domiciliary application once a day for 15 days after the visits (no rinsing and eating for 30 minutes after mouthwash application).
  Arms: Control Group

SUMMARY:
This is a randomized controlled clinical trial (RCT). After signing the informed consent, patients satisfying the inclusion criteria will undergo supragingival and subgingival professional oral hygiene of both arches performed with ultrasonic instrumentation with PEEK inserts, manual instrumentation with PEEK curettes and air polishing with glycine powder.

After that, the sample will be randomly divided into 2 groups based on the domiciliary assigned treatment:

* Aftoral® Oral Gel solution with Hyaluronic Acid, Xylitol and glycerophosphoinositol for the domiciliary use for 15 days for 2 peri-implant mucositis sites.
* Unidea® Chlorhexidine digluconate Mouthwash 0,20% administration for the domiciliary application for 15 days for 2 peri-implant sites.

The study will last 6 months. Patients will be visited at: T0, after 1 month from T0 (T1), after 3 months (T2), after 6 months (T3), after 9 months (T4) and after 12 months (T5). Professional hygiene will be performed again at T3.

At each recall session were collected a satisfaction questionnaire of the products (taste, smell, consistency, persistence and ease of application) and the following periodontal clinical indices, using a PEEK probe on each peri-implant site:

* conditions of the marginal mucosa (swelling and erythema),
* migration of the marginal mucosa,
* PPD (Probing Pocket Depth),
* BOP% (Bleeding on Probing),
* BS (Bleeding Score),
* Suppuration,
* PCR% (Plaque Control Record),

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial (RCT). 60 patients are expected to be enrolled. After signing the informed consent, patients satisfying the inclusion criteria will undergo supragingival and subgingival professional oral hygiene of both arches performed with ultrasonic instrumentation with PEEK inserts, manual instrumentation with PEEK curettes and air polishing with glycine powder.

After that, the sample will be randomly divided into 2 groups based on the domiciliary assigned treatment:

* Aftoral® Oral Gel solution with Hyaluronic Acid, Xylitol and glycerophosphoinositol for the domiciliary use for 15 days for 2 peri-implant mucositis sites.
* Unidea® Chlorhexidine digluconate Mouthwash 0,20% administration for the domiciliary application for 15 days for 2 peri-implant sites.

The study will last 6 months. Patients will be visited at: T0, after 1 month from T0 (T1), after 3 months (T2), after 6 months (T3), after 9 months (T4) and after 12 months (T5).

At T3, professional hygiene will be performed again.

At each recall session were collected a satisfaction questionnaire of the products (taste, smell, consistency, persistence and ease of application) and the following periodontal clinical indices, using a PEEK probe on each peri-implant site:

* conditions of the marginal mucosa (swelling and erythema),
* Marginal mucosal condition,
* PPD (Probing Pocket Depth),
* BOP% (Bleeding on Probing),
* BS (Bleeding Score),
* Suppuration,
* PCR% (Plaque Control Record).

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years
* presence of at least one site suffering from peri-implant mucositis with PPD > or equal to 5 mm
* no systemic, metabolic and autoimmune disease
* compliant patients

Exclusion Criteria:

* absence of dental implants
* neurologic, psychiatric and mental diseases
* patients taking bisphosphonates in the last 12 months
* patients taking antibiotics during the study
* pregnant and breastfeeding women
* patients undergoing anticancer treatment
* allergy to chlorhexidine or hyaluronic acid
* sites with peri-implantitis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Change in Probing Depth (PD) | Baseline (T0), after 1 (T1), 3 (T2), 6 (T3), 9 (T4) and 12 months (T5)
  Evaluation (in mm) of the depth of the gingival sulcus, through a millimeter periodontal PEEK probe; it is detected from the gingival margin to the bottom of the gingival sulcus or periodontal pocket, evaluated at 6 sites.
Change in Bleeding on Probing (BOP%) | Baseline (T0), after 1 (T1), 3 (T2), 6 (T3), 9 (T4) and 12 months (T5)
  Quantitative assessment (percentage) of the bleeding sites (6 per tooth in total).
  Formula = n ° bleeding sites / n ° probed sites x100
Change in Bleeding Score (BS - Mombelli et al.) | Baseline (T0), after 1 (T1), 3 (T2), 6 (T3), 9 (T4) and 12 months (T5)
  Scoring criteria:
  0: no bleeding
  1. isolated visible spots
  2. blood forms a confluent red line on the mucosal margin
  3. profuse and copious bleeding
Change in Plaque Control Record (PCR%) | Baseline (T0), after 1 (T1), 3 (T2), 6 (T3), 9 (T4) and 12 months (T5)
  Evaluation of the presence of plaque on the 4 surfaces of teeth on the total amount of dental surfaces.
  Formula = n ° sites with plaque / total n ° of dental surfaces x100
Change in marginal mucosa condition | Baseline (T0), after 1 (T1), 3 (T2), 6 (T3), 9 (T4) and 12 months (T5)
  Scoring criteria:
  0: normal mucosa
  1. minimal inflammation with color change and minor edema
  2. moderate inflammation with redness, edema and glazing
  3. severe inflammation with redness, edema, ulceration and spontaneous bleeding without probing
Change in Suppuration (%) | Baseline (T0), after 1 (T1), 3 (T2), 6 (T3), 9 (T4) and 12 months (T5)
  Dichotomous scoring (yes/no) of suppurating sites

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, MS, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the Principal Investigator.